CLINICAL TRIAL: NCT07018401
Title: Pomalidomide for the Treatment of Bleeding in Hereditary Hemorrhagic Telangiectasia After Trial Longitudinal Assessment Study (PATH-HHT ATLAS)
Brief Title: Pomalidomide for the Treatment of Bleeding in Hereditary Hemorrhagic Telangiectasia Longitudinal Assessment Study
Acronym: PATH-HHT ATLAS
Status: Active, not recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: The Cleveland Clinic (Other); University of North Carolina, Chapel Hill (Other); University of California, San Francisco (Other); Mayo Clinic (Other); University of Utah (Other); University of California, San Diego (Other); University of Florida (Other); Medical College of Wisconsin (Other); Johns Hopkins University (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Hanny Al-Samkari, MD, Classical Hematologist, Clinical Investigator, Massachusetts General Hospital
Other Study IDs: InHIBIT-002
Record Dates: First submitted 2025-05-28; First posted 2025-06-12 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-06

CONDITIONS: Hereditary Hemorrhagic Telangiectasia (HHT)
Keywords: hereditary hemorrhagic telangiectasia; HHT; Osler-Weber-Rendu; pomalidomide; PATH-HHT; PATH-HHT ATLAS
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic | interventions — pomalidomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Pomalidomide — Oral pomalidomide up to 4 mg daily
  Other Names: Pomalyst

SUMMARY:
This is a multicenter U.S. longitudinal study evaluating patients with hereditary hemorrhagic telangiectasia who participated in the PATH-HHT clinical trial of pomalidomide for the treatment of HHT. This study is a longitudinal assessment of safety and effectiveness of pomalidomide in HHT in clinical trial participants following completion of the double-blind, placebo-controlled study.

DETAILED DESCRIPTION:
Hereditary Hemorrhagic Telangiectasia (HHT) is an autosomal dominant condition characterized by disordered angiogenesis that affects 1 in 5,000 people. It results in numerous clinical complications including severe recurrent epistaxis, gastrointestinal bleeding, chronic iron deficiency anemia (and possible transfusion dependence), high-output cardiac failure, and many others. In recognition that elevated levels of vascular endothelial growth factor (VEGF) are elevated in HHT, anti-angiogenic drugs are now being used to treat HHT off-label to manage HHT-associated bleeding. A primary agent used for this purpose is pomalidomide, an oral immunomodulatory drug with antiangiogenic properties. Pomalidomide was demonstrated to be efficacious over a 6-month treatment period in the multicenter U.S. randomized controlled PATH-HHT Study. The present study is the successor to PATH-HHT, the PATH-HHT ATLAS (After Trial Longitudinal Assessment Study). This study will evaluate the long-term impact of pomalidomide on epistaxis (as measured by the validated ESS, epistaxis severity score), gastrointestinal bleeding, and iron deficiency anemia (as assessed by hemoglobin measurements, red blood cell transfusions, and intravenous iron infusions).

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis of HHT as defined by the Curacao criteria
2. Age > 18 years
3. Platelet count ≥ 100 x 109/L prior to pomalidomide initiation
4. WBC ≥ 2.5 x 109/L prior to pomalidomide initiation
5. INR ≤ 1.4 and normal ± 2 sec activated partial thromboplastin time (aPTT) by local laboratory criteria (except for patients on a stable dose of warfarin or direct oral anticoagulants)
6. Epistaxis severity score ≥ 3 measured over the preceding month
7. A requirement for anemia, as determined by local laboratory normal ranges, and/or parenteral infusion of at least 250 mg of iron or transfusion of 1 unit of blood over the 24 weeks preceding the screening visit
8. All study participants must agree to be registered into the FDA mandated POMALYST REMS program, and be willing and able to comply with the requirements of the POMALYST REMS program
9. Females of childbearing potential (FCBP)† must adhere to the pregnancy testing schedule mandated by the POMALYST REMS program
10. Prior enrollment on PATH-HHT study (NCT03910244)

    * A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Exclusion Criteria:

1. Women currently breast feeding or pregnant
2. Renal insufficiency, serum creatinine > 2.0 mg/dl
3. Hepatic insufficiency, bilirubin > 2.0 (or >4.0 in the setting of a prior clinical or genetic diagnosis of Gilbert's syndrome) or transaminases > 3.0x normal
4. Prior treatment with thalidomide or other non-pomalidomide immunomodulatory imide drugs (IMiDs) within previous 6 months
5. Prior treatment with bevacizumab (systemic or nasal) within previous 6 weeks
6. Prior treatment with pazopanib within previous 6 weeks
7. The use of octreotide or estrogens within the previous month
8. History of prior unprovoked thromboembolism confirmed by venous ultrasound or other imaging modalities
9. Known peripheral neuropathy, confirmed by neurologic consultation
10. Known underlying hypoproliferative anemia (i.e. myelodysplasia, aplastic anemia)
11. Currently enrolled in other drug trials
12. Known hypersensitivity to thalidomide or lenalidomide
13. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
14. Known SMAD-4 mutation, unless there has been a colonoscopy with normal (negative) results, or in which the patient has had no more than 5 small (in the opinion of the gastroenterologist) colonic polyps completely removed within the preceding 18 months
15. Anything that in the investigator's opinion is likely to interfere with completion of the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with hereditary hemorrhagic telangiectasia and moderate-to-severe bleeding who previously enrolled in the PATH-HHT trial
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Epistaxis Severity Score | 12 months
  Validated bleeding scale in HHT scored between 0-10, higher scores indicate worse bleeding

SECONDARY OUTCOMES:
Serum hemoglobin (g/dL) | 12 months
Hematologic Support Score | 12 months
  Composite hematologic endpoint, higher scores indicate more hematologic support requirements
Intravenous iron infusion (mg elemental iron) | 12 months
Red cell transfusion (units of packed red blood cells) | 12 months
Incidence of treatment-emergent adverse events (safety) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Zhang, MD, Study Director — Stanford University
Locations (11):
- United States (11):
  - University of California-San Diego, San Diego, California
  - University of California-San Francisco, San Francisco, California
  - University of Florida, Gainesville, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of North Carolina, Chapel HIll, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang E, Kasthuri RS, Parambil J, Prasad V, Iyer V, Whitehead K, Hodges PG, Pishko A, Conrad M, Phelan D, Rodriguez-Lopez J, McCrae KR, Al-Samkari H. Pomalidomide for Hereditary Hemorrhagic Telangiectasia: After Trial Longitudinal Assessment Study (PATH-HHT ATLAS). Blood Adv. 2026 Jan 9:bloodadvances.2025018382. doi: 10.1182/bloodadvances.2025018382. Online ahead of print. PMID 41512167